CLINICAL TRIAL: NCT04639271
Title: A Single-arm, Open-label Study Of Pyrotinib Combined WithTrastuzumab And Abraxane in Patients With Brain Metastases From HER2-positive Metastatic Breast Cancer
Brief Title: Pyrotinib, Trastuzumab And Abraxane in HER2-positive MBC With Brain Metastasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Zhiyong Yu, Principal Investigator, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ShandongCHI-16
Record Dates: First submitted 2020-11-19; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer; HER2-positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; Trastuzumab; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pyrotinib Plus Trastuzumab And Abraxane (Experimental): Pyrotinib Plus Trastuzumab And Abraxane
  Interventions: Drug: Pyrotinib Plus And; Drug: Trastuzumab; Drug: Abraxane

INTERVENTIONS:
Drug: Pyrotinib Plus And — Pyrotinib::400mg/d,qd,po
Drug: Trastuzumab — 8 mg/kg intravenously (IV) on Day 1 of Cycle 1, followed by 6 mg/kg on Day1 of each 21-day cycle
Drug: Abraxane — Abraxane 125mg/M2, qw iv

SUMMARY:
The purpose of this study is to assess the efficacy and safety of pyrotinib combined with trastuzumab and abraxane in HER2-positive MBC with brain metastasis.

DETAILED DESCRIPTION:
Overexpression of HER2 is associated with increased incidence of brain metastases in breast cancer, accounting for about 20-50% of HER2 positive breast cancer. Treatment strategy ranged from local therapies to systemic anti-HER2 therapies, prognosis of patients with brain metastases remains poor. Previous clinical trials had demonstrated the efficacy of trastuzumab and TKIs for brain metastasis.

Pyrotinib is an oral tyrosine kinase inhibitor targeting both HER-1 and HER-2 receptors. We designed the study to explore the efficacy and safety of pyrotinib combined with trastuzumab and abraxane in HER2-positive MBC with brain metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18 years.
* ECOG performance status ≤2.
* Histologically or cytologic confirmed HER2 positive advanced breast cancer.
* MRI confirmed brain metastases. According to RECIST 1.1, at least one measurable lesion exists.
* No limit of previous chemotherapy lines.
* Previously have not reveived capecitabine or disease progression of capecitabine after 6 months, or progression of capecitabine adjuvant therapy after one year;
* Life expectancy of more than 3 months.
* Required laboratory values including following parameters: ANC: ≥ 1.5 x 10^9/L;Platelet count: ≥ 100 x 10^9/L;Hemoglobin: ≥ 9.0 g/dL;Total bilirubin: ≤ 1.5 x upper limit of normal (ULN);ALT and AST: ≤ 1.5 x ULN (or ≤ 5×ULN in patients with liver metastases);BUN and creatine clearance rate: ≥ 50 mL/min;LVEF: ≥ 50%;QTcF: < 470 ms for female and < 450 ms for male.
* Signed the informed consent form prior to patient entry.

Exclusion Criteria:

* Patients with brain metastases who have extensive meningeal metastases and are treated with hormone dehydration.
* Subjects with third space fluid(such as a large amount of pleural effusion and ascites) that can not be controled by drainage or other methods. (such as pleural effusion and ascites).
* Received whole brain radiotherapy, chemotherapy, surgery or target therapy within 2 weeks prior to randomization. Received hormone therapy within 1 weeks prior to randomization, Received the nitrosoureas or mitomycin chemotherapy within 6 weeks prior to randomization.
* Participated in other clinical trial within 4 weeks prior to randomization.
* Treated or treating with HER2 tyrosine kinase inhibitors (TKIs) (including Lapatinib, Neratinib and Pyrotinib).
* Second malignancies within 5 years, except for cured carcinoma in-situ of uterine cervix, skin basal cell carcinomaand squamous-cell carcinoma.
* Receiving any other anti-tumor therapies at time of study screening visit.
* There are no other serious and/or uncontrolled diseases that may affect research participation, including any of the following: (1) unable to swallow, chronic diarrhea and intestinal obstruction and factors influencing the usage of oral administration; (2) has allergies or a known history of hypersensitivity to the drug components of this program; History of Immunodeficiency, acquired or congenital immunodeficiency (HIV positive) ,history of organ transplantation; (3) History of any kind of Heart disease, including 1) Myocardial infarction; 2) Heart failure; 3) Any other heart disease judged by researcher as not suitable for participating in this study, etc; (4) Infection.
* All female patients in breastfeeding period or in child-bearing period or with positive pregnancy test result or refusing to take a reliable method of birth control during the study.
* Any other situations judged by investigator as not suitable for participating in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) of Intracranial Lesion | Estimated up to 1 year
  Refers to the proportion of patients whose Intracranial Lesion have shrunk to a certain proportion and maintained for a certain period of time, including cases of CR and PR, RECIST 1.1 were used to assess objective tumor remission
Progression Free Survival(PFS) of Intracranial Lesion | Estimated up to 1 year
  the date from the first dose to the first occurrence of Intracranial Lesion progression or death from any cause, whichever occurs first

SECONDARY OUTCOMES:
Progression Free Survival(PFS) | Estimated up to 1 year
  the date from the first dose to the first occurrence of disease progression or death from any cause, whichever occurs first
Objective Response Rate (ORR) | Estimated up to 1 year
  Refers to the proportion of patients whose lesion have shrunk to a certain proportion and maintained for a certain period of time, including cases of CR and PR, RECIST 1.1 were used to assess objective tumor remission
disease control rate(DCR) | Estimated up to 1 year
  Percentage of confirmed complete remission (CR), partial remission (PR), and disease stable (SD) cases in patients with evaluable efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- Zhiyong Yu, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No